CLINICAL TRIAL: NCT03732027
Title: Anterior Abdominal Blocks for Postoperative Pain Control in Obese Patients Undergoing Major Gynecological Surgery: Surgical Transversus Abdominis Plane Block Versus Surgical Rectus Sheath Block
Brief Title: Anterior Abdominal Blocks for Postoperative Pain Control in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Khairy Elbeialy, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R55 /2018
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Block [TB] group (Active Comparator): Patients will receive Surgical Transversus Abdominis Plane Block
  Interventions: Procedure: Surgical Transversus Abdominis Plane Block
- Rectus Sheath Block [RB] group (Active Comparator): Patients will receive Surgical Rectus Sheath Block
  Interventions: Procedure: Surgical Rectus Sheath Block

INTERVENTIONS:
Procedure: Surgical Transversus Abdominis Plane Block — At the end of operation and after hemostasis, 20 ml of 0.25% bupivacaine will be injected intra-abdominally into the Transversus Abdominis plane at the midpoint of the line connecting the crista iliaca and inferior costal margin and at two locations in the lateral abdominal wall at 3-4 cm inferior to the previous midline injection. The same procedure will be repeated on the opposite side using an identical amount of local anesthetic.
  Arms: Transversus Abdominis Block [TB] group
Procedure: Surgical Rectus Sheath Block — At the end of operation and after hemostasis,20 ml 0.25% bupivacaine will be administered slowly under direct vision after careful aspiration to the rectus sheath space which is present inbetween rectus abdominis muscle and the posterior layer of its sheath at the upper pole of the midline incision by time of closure of the anterior abdominal wall. The procedure will be repeated on the opposite side.
  Arms: Rectus Sheath Block [RB] group

SUMMARY:
The purpose of this study is to compare between two surgical techniques for anterior abdominal wall blocks in obese patients Undergoing Major Gynecological Surgery: Surgical Transversus Abdominis Plane [TAP] block versus Rectus Sheath block as regards the efficacy and adverse effects

ELIGIBILITY:
Inclusion Criteria:

* female patients
* undergoing major gynecological surgery with supraumbilical midline incision the first time
* Body mass index (BMI) more than 40.

Exclusion Criteria:

* patient refusal to participate in the study,
* reoperation,
* addiction
* alcohol abuse
* hypersensitivity or allergy to the study drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine consumption | First 24 hours postoperatively

SECONDARY OUTCOMES:
Numerical rate scale | First 24 hours postoperatively
  Postoperative pain will be assessed at rest and coughing using numerical rate scale (NRS) patients are asked to rate their pain on a scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain possible,".
Postoperative respiratory functions | First 24 hours postoperatively
  will be measured using incentive spirometer. Patients were asked to do sustained maximal inspiration (SMI) three times. Then average SMI will be recorded. They will be instructed prior to induction of general anesthesia about the usage of incentive spirometer then a basal measurement will be obtained. After recovery, measurement will be obtained on 60 min, 6 hours, 12 hrs and 24 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa AK Elbeialy, MD, Principal Investigator — Faculty of Medicine,Ain Shams University
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided